CLINICAL TRIAL: NCT06081621
Title: A Multi-center, Randomized, Double-Blinded, Parallel and Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of REGEND001 Cell Therapy in Idiopathic Pulmonary Fibrosis (IPF) Patients
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of REGEND001 Cell Therapy on Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regend Therapeutics (Industry)
Collaborators: Peking Union Medical College Hospital (Other); RenJi Hospital (Other); Ruijin Hospital (Other); The Second Affiliated Hospital of Xiamen Medical College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REGEND001-IPF-231-V1.3
Record Dates: First submitted 2023-09-17; First posted 2023-10-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REGEND001 (Experimental)
  Interventions: Biological: REGEND001
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: REGEND001 — REGEND001: 1-1.5×10^6 bronchial basal cells/kg administrated by bronchoscopy.
  Arms: REGEND001
Biological: Placebo — Placebo: Sodium chloride injection administrated by bronchoscopy.
  Arms: Placebo

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a serious chronic (long term) disease with injury of lung tissues. REGEND001 is a cell therapy product, made from bronchial basal cells with ability to regenerate lung tissue, is promising to IPF treatment. This is a multi-center, randomized, double-blinded, parallel and placebo-controlled phase II clinical study to evaluate the efficacy and safety of REGEND001 in IPF patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 40 to 75;
* Subjects diagnosed with IPF according to guidelines for the diagnosis of idiopathic pulmonary fibrosis 2022 edition;
* Subjects with DLCO (measured/predicted value) ≥30% and <80%, and FVC (measured/predicted value) ≥50% within 3 months prior to screening
* Subjects tolerant to bronchofiberscope;
* Subjects tolerant to test of lung function;
* Subjects able to voluntarily sign the informed consent and cooperate with the completion of pulmonary function tests;

Exclusion Criteria:

* Female subject who is pregnant, nursing, or planning to be pregnant in half a year after using this product (or male subjects planning to have a pregnant spouse);
* At the time of screening, subject who is positive in each of treponema pallidum antibody (TP-Ab), human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody test, except the following: (1) Hepatitis B virus carriers (only HBsAg positive, no hepatitis symptoms and signs, all liver function tests are normal); (2) Cured hepatitis C patients with negative result in HCV ribonucleic acid (RNA) test.
* Subject with malignant tumors or a history of malignant tumors;
* Subject with severe anemia, poorly controlled agranulocytosis and thrombocytopenia at screening;
* Subject at risk of suicide or has a history of mental illness or epilepsy at the time of screening;
* Subject with severe arrhythmias or atrioventricular block of degree II or above, shown by 12-lead Electrocardiogram (ECG);
* Subject who participated in other interventional clinical trials in the past 3 months;
* Subject assessed as inappropriate to participate in this clinical trial by investigators.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Comparison of the area under the curve (AUC) of DLCO measured values at each visit from baseline to week 24 between the REGEND001 group and the placebo group. | 12 and 24 weeks after treatment
  DLCO is measured by the single-breath method. Improvement is defined as an increase in DLCO from baseline.

SECONDARY OUTCOMES:
Change from baseline in lung diffusing capacity | 12 and 24 weeks after treatment
  DLCO will be used to evaluate the lung diffusing capacity. DLCO test refers to the diffusing capacity for carbon monoxide in the lungs. It's a type of pulmonary function test that helps to assess how well gas is exchanged between the lungs and the bloodstream.

OTHER OUTCOMES:
Change from baseline in lung ventilatory capacity | 12 and 24 weeks after treatment
  Forced vital capacity (FVC) and forced expiratory volume in one second (FEV1) will be used to evaluate the lung ventilatory capacity. FVC indicates the volume of air that can forcibly be blown out after full inspiration. FEV1 is the volume of breath exhaled with effort in one second.
Progression-free survival (PFS) | Within 24 weeks after treatment
  PFS refers to the time from randomization or initiation of treatment to the occurrence of disease progression or death.
Change from baseline in St. George's respiratory questionnaire (SGRQ) scale | 12 and 24 weeks after treatment
  Quality of life was assessed by St. George's respiratory questionnaire (SGRQ) scale. Total score, ranged from 0 to 100, is the sum of points from all items. A higher value represents a worse outcome.
Change from baseline in 6-minute-walk test (6MWT) | 12 and 24 weeks after treatment
  The 6MWT is a commonly used test for the objective assessment of functional exercise capacity by testing the distance patients can walk at the fastest speed within 6 minutes.
Time from enrollment to all-cause death | up to 24 weeks(first period), 5 years (second period).
  Time from enrollment to all-cause death is used to evaluate the overall survival of the population.
Blood oxygen saturation | 12 and 24 weeks after treatment
  Blood oxygen saturation is the measure of how much oxygen is traveling through body in red blood cells.
Change from baseline in images of lung by high resolution computed tomography (HR-CT) | 12 and 24 weeks after treatment
  HR-CT images of lung will be analyzed to indicate the change of pulmonary structure.
Change from baseline in C-reactive protein (CRP) | 12 and 24 weeks after treatment
  The level of CRP increases when there's inflammation in the body.
Time to acute exacerbations of idiopathic pulmonary fibrosis (AE-IPF) | Within 24 weeks after treatment
  AE-IPF is an often deadly complication of IPF, which is defined as an acute, clinically significant respiratory deterioration characterized by evidence of new widespread alveolar abnormality.
Temperature | Within 24 weeks after treatment
  Number of cases with abnormal body temperature.
Breathing | Within 24 weeks after treatment
  Number of cases with abnormal breathing.
Pulse | Within 24 weeks after treatment
  Number of cases with abnormal pulse.
Blood pressure | Within 24 weeks after treatment
  Number of cases with abnormal blood pressure.
Symptoms, physical examination | Within 24 weeks after treatment
  Number of cases with abnormal physical examination
12-lead ECG | Within 24 weeks after treatment
  Number of cases with abnormal 12-lead Electrocardiogram (ECG).
Blood routine | Within 24 weeks after treatment
  Number of cases with abnormal laboratory test results
Liver & Kidney function check | Within 24 weeks after treatment
  Number of cases with abnormal results in Liver & Kidney function check
Blood sugar | Within 24 weeks after treatment
  Number of cases with abnormal results
Function of blood clotting | Within 24 weeks after treatment
  Number of cases with abnormal function of blood clotting.
Antibody testing for autoimmune diseases | Within 24 weeks after treatment
  Antibodies related to autoimmune diseases are tested for safety assessment
Carcinoembryonic antigen (CEA) | Within 24 weeks after treatment
  CEA is a tumor marker used for early diagnosis of lung cancer.Clinically significant changes of this markers will be assessed.
Neuron-specific enolase (NSE) | Within 24 weeks after treatment
  NSE is a tumor marker significantly elevated in small cell lung cancer. Clinically significant changes of this marker will be assessed
Cytokeratin-19-fragment (CYFRA21-1) | Within 24 weeks after treatment
  CYFRA21-1 is a tumor marker which is valuable for the pathological classification and prognosis evaluation of lung cancer. Clinically significant changes of this marker will be assessed
Squamous cell carcinoma antigen (SCC) | Within 24 weeks after treatment
  SCC is a specific marker for lung squamous cell carcinoma. Clinically significant changes of this marker will be assessed
Other cases of adverse effects | Within 24 weeks after treatment
  Other cases of adverse effects will be recorded and compared.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - Ruijin Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No